CLINICAL TRIAL: NCT05690399
Title: Evaluation of Clinical and Pathological Characteristics and Routine Treatment of Patients With Prostate Cancer in 2 Centers in Asyut
Brief Title: Evaluation of Clinical and Pathological Characteristics and Routine Treatment of Patients With Prostate Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aml Mohamed Haridy, Evaluation of clinical and pathological characteristics and routine treatment of patients with prostate cancer in 2 centers in Asyut, Assiut University
Other Study IDs: Prostate cancer
Record Dates: First submitted 2023-01-10; First posted 2023-01-19 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Radiotherapy — Effect of radiotherapy on patients

SUMMARY:
To evaluate clinical and pathological characteristics and treatment protocol and outcomes of patients with prostate cancer in 2 centers of Asyut from 2013 to 2023

DETAILED DESCRIPTION:
Inclusion criteria :

* Male patient , Age ≥ 40 yo
* Diagnosed as prostate cancer from ( 2013- 2023 ) proved by biopsy in South Egypt Cancer Institute "SECI" & Asyut clinical oncology department
* Newly diagnosed/ metastatic at presentation
* ECOG 0-4

  • Exclusion criteria:
* Having Other types of malignancy.

ELIGIBILITY:
Inclusion Criteria:

* Male patient , Age ≥ 40 yo
* Diagnosed as prostate cancer from ( 2013- 2023 ) proved by biopsy
* Newly diagnosed/ metastatic at presentation
* ECOG 0-4

Exclusion Criteria:

* Having Other types of malignancy.

Min Age: 40 Years | Sex: Male
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Diagnosed as prostate cancer from ( 2013- 2023 ) proved by biopsy
  - Newly diagnosed/ metastatic at presentation
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Clinical and pathological characteristics and routine treatment of patients with prostate cancer in 2 centers in Asyut in previous 10 years | Baseline
  Clinical and pathological characteristics and routine treatment of patients with prostate cancer in 2 centers in Asyut in previous 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Assiut University, Principal Investigator — Assiut University

REFERENCES:
- See also: Cancer Stat Facts: Prostate Cancer [Internet]. SEER, 2018. — http://seer.cancer.gov/statfacts/html/prost.html
- See also: M Alizadeh, S Alizadeh, Glob J Health Sci, 6: 2014. Survey of clinical and pathological characteristics and outcomes of patients with prostate cancer — http://www.ccsenet.org/journal/index.php/gjhs/article/view/38296